CLINICAL TRIAL: NCT05417893
Title: To Compare the Safety and Performance of MeRes100 Sirolimus Eluting BioResorbable Vascular Scaffold System Versus Contemporary DES Platforms in Patients With de Novo Coronary Artery Lesions
Brief Title: Non-inferiority Clinical Trial to Compare the Safety and Performance of MeRes100 Sirolimus-eluting BioResorbable Vascular Scaffold System Versus Contemporary DES Platforms in Patients With de Novo Coronary Artery Lesions
Acronym: MeRethonRCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLS/MER/MeRethon RCT
Record Dates: First submitted 2022-03-07; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort-1: MeRes 100 BRS (Active Comparator): 1248 subjects will be delivered with MeRes 100 BRS
  Interventions: Device: MeRes 100 Sirolimus-eluting Bioresorbable Vascular Scaffold System (BRS)
- Cohort- 2: Contemporary DES platforms (Active Comparator): 624 subjects will be delivered with Contemporary DES
  Interventions: Device: MeRes 100 Sirolimus-eluting Bioresorbable Vascular Scaffold System (BRS)

INTERVENTIONS:
Device: MeRes 100 Sirolimus-eluting Bioresorbable Vascular Scaffold System (BRS) — The MeRes100™ BRS (Meril Life Sciences Pvt. Ltd., India) is a novel thin-strut second-generation sirolimus-eluting poly-L-lactic acid (PLLA)-based bioresorbable coronary scaffold. The first-in-human MeRes-1 trial demonstrated the safety and effectiveness of MeRes100 BRS in the treatment of de novo coronary lesions with lower major adverse cardiac events (MACE) rate (0.93%) and notably, the absence of scaffold thrombosis at one-year follow-up. MeRes100 sirolimus-eluting bioresorbable vascular scaffold system is expected to bioresorb in the artery, approximately over a period of three years and thus, preventing chance of late clinical events like late scaffold thrombosis rates. The imaging analysis has shown that in-segment late lumen loss and in-scaffold late lumen loss (LLL) did not change significantly at two years follow-up as compared to six months data.
  Other Names: XIENCE family Everolimus-eluting Coronary Stent System (EES); Resolute Zotarolimus-eluting Coronary Stent System (ZES); Synergy EES; BioMime/Metafor/Proficient family Sirolimus-eluting Coronary Stent System (SES)

SUMMARY:
This is a prospective, open-label, multicentre, randomized, non-inferiority clinical trial to compare the safety and performance of MeRes100 Sirolimus-eluting BioResorbable Vascular Scaffold System versus Contemporary drug-eluting stent platforms in patients with de novo coronary artery lesions at 60 investigational sites globally (including India).

The primary objective of this study is to evaluate safety and performance of MeRes100 BRS in comparison with XIENCE family EES/Resolute ZES/Synergy EES/BioMime/Metafor/Proficient family SES in patients with de novo coronary artery lesions with reference vessel diameter of ≥2.75 mm to ≤4.0 mm and lesion length ≤34 mm.

Subject's Clinical/Telephonic Follow-up will be taken at [Time Frame: 30 days (± 7 days) clinical follow-up, 6 month (± 28 days) clinical follow-up, 1 year (± 28 days) clinical follow-up, 2 years (± 28 days) telephonic follow-up, 3 years (± 28 days) clinical follow-up, 4 years (± 28 days) telephonic follow-up and 5 years (± 28 days) clinical follow-up]

DETAILED DESCRIPTION:
This is a prospective, open-label, multicentre, randomized, non-inferiority clinical trial to compare the safety and performance of MeRes100 Sirolimus-eluting BioResorbable Vascular Scaffold System versus Contemporary drug-eluting stent platforms in patients with de novo coronary artery lesions at 60 investigational sites globally (including India).

The primary objective of this study is to evaluate safety and performance of MeRes100 BRS in comparison with XIENCE family EES/Resolute ZES/Synergy EES/BioMime/Metafor/Proficient family SES in patients with de novo coronary artery lesions with reference vessel diameter of ≥2.75 mm to ≤4.0 mm and lesion length ≤34 mm.

The MeRes100™ BRS (Meril Life Sciences Pvt. Ltd., India) is a novel thin-strut second-generation sirolimus-eluting poly-L-lactic acid (PLLA)-based bioresorbable coronary scaffold is indicated for improving coronary luminal diameter in patients with symptomatic ischemic heart disease due to de novo lesion in native coronary arteries in patients eligible for percutaneous transluminal coronary angioplasty and scaffolding procedures.

After informed consent provided by the subject and confirmation of eligibility criteria and diagnostic angiography, subject will be randomized (2:1) to MeRes100 BRS or Contemporary DES using centralized web-based system.

Subject's Clinical/Telephonic Follow-up will be taken at [Time Frame: 30 days (± 7 days) clinical follow-up, 6 month (± 28 days) clinical follow-up, 1 year (± 28 days) clinical follow-up, 2 years (± 28 days) telephonic follow-up, 3 years (± 28 days) clinical follow-up, 4 years (± 28 days) telephonic follow-up and 5 years (± 28 days) clinical follow-up]

ELIGIBILITY:
General Inclusion Criteria:

1. Male or female subject ≥18 years of age
2. Subject who has provided written informed consent
3. Subject must agree to undergo all clinical investigations and follow-up visits as per protocol
4. Subject with documented myocardial ischemia (e.g. stable, unstable angina, or silent ischemia) and who are eligible candidates for elective percutaneous coronary intervention (PCI)
5. Subject must agree not to participate in any other clinical trial for a period of one year following the index procedure. This includes clinical trials of medications and/or invasive procedures. Questionnaire-based studies, or other studies that are non-invasive and do not require medication are allowed

Angiographic Inclusion Criteria:

1. One de novo target lesion or up-to two de novo target lesions in different epicardial vessels: Different epicardial vessels are defined as left anterior descending artery (LAD) and its branches, left circumflex artery (LCX) arteries and its branches, and right coronary arteries (RCA) and its branches. Thus, for example, the subject must not have two target lesions required to be treated at the LAD and its branches at the same time
2. Each target lesion can be fully covered by one scaffold
3. Target lesion with angiographic evidence of ≥70% stenosis (by visual estimation) and ≥50% (by QCA estimation) with TIMI flow of ≥1. If the target lesion is <70% stenosed, there must be an evidence of ischemia as per ECG or nuclear scan or fractional flow reserve (FFR)
4. Target lesion(s) located in native coronary artery with reference vessel diameter (RVD) of ≥2.75 mm to ≤4.0 mm and length ≤34 mm by QCA or by visual estimation

Exclusion Criteria:

1. Known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, antiplatelet medication specified for use in the study (clopidogrel, prasugrel, ticlopidine inclusive), everolimus, sirolimus or its analog or derivative, poly (L-lactide), poly (DL-lactide), cobalt, PLGA [poly(DL-lactide-co-glycolide)], chromium, nickel, tungsten, stainless steel, platinum, platinum-chromium alloy, iron, molybdenum, amorphous silicon carbide, acrylic and fluoropolymers or contrast sensitivity that cannot be adequately pre-medicated
2. Any PCI <6 months prior to the index procedure
3. Previous CABG or PCI in the target vessel(s)
4. Left ventricular ejection fraction (LVEF) <30% as evaluated by any non-invasive imaging method including but not limited to, echocardiogram, angiography, Magnetic Resonance Imaging (MRI), Multiple-Gated Acquisition (MUGA) scan, radionuclide ventriculography, Positron Emission Tomography (PET) scan, etc. For subjects with stable Coronary Artery Disease (CAD), LVEF may be obtained within 6 months prior to the procedure. For Acute coronary syndrome (ACS) subjects, LVEF must be evaluated during hospitalization or during index procedure but prior to randomization for confirming the subject's eligibility.
5. Concurrent medical condition with less than three years of life expectancy
6. Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months of baseline visit
7. Renal insufficiency as estimated by Glomerular Filtration Rate (GFR) <30 ml/min/1.73m2 or dialysis at the time of screening or creatinine level is more than 1.5 mg/dl
8. Subject with cardiac arrhythmia detected at the time of screening
9. Subject is on immunosuppressant therapy and has immunosuppressive or autoimmune disease.
10. Subject with hepatic disorder or chronic liver disease, known aplastic anaemia, platelet count <100,000 cells/mm3 or > 700,000 cells/mm3, a WBC of < 3,000 cells/mm3
11. Subject with prior brachytherapy of the target lesion or use of brachytherapy for the treated site restenosis
12. Subject has a history of bleeding diathesis or coagulatory disease, refuses blood transfusion, significant gastrointestinal or urinary bleed within the past 12 months
13. Subject who underwent or needs organ transplant
14. Planned PCI for any clinically significant lesion after index procedure
15. Planned surgery within 12 months after index procedure
16. Pregnant or nursing subject and those who plan pregnancy in the period until 5 years following index procedure (Female subject of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure and contraception must be used during participation in this trial)
17. Any newly onset acute myocardial infarction within 1 week (<7days) or, myocardial enzyme has not returned to normal level (clinically non-significant) after myocardial infarction.
18. Subject with significant peripheral vascular disease that precludes safe access to sheath or catheter

Angiographic Exclusion Criteria:

1. Target lesion located within 3 mm of the origin of the LAD or LCx
2. Target lesion involving a bifurcation lesion with side branch ≥2 mm in diameter
3. Highly calcified lesions Classification of calcification: moderate calcification - discontinuous dotted high density image; severe calcification - continuous high density image around the whole vessel wall under continuous X ray by multiple positions.
4. Target lesion which prevents complete balloon pre-dilatation, defined as full balloon expansion with the following outcomes:

   1. Residual % Diameter Stenosis (DS) is < 40% (per visual estimation), (≤ 20% is strongly recommended).
   2. TIMI Grade-3 flow (per visual estimation).
   3. No angiographic complications (e.g., no-reflow, distal embolization, side branch closure).
   4. No dissections NHLBI grade D-F.
   5. No chest pain lasting > 5 minutes.
   6. No ST depression or elevation lasting > 5 minutes
5. Total occlusion (TIMI flow 0), prior to wire crossing
6. Excessive tortuosity (≥ two 45° angles), or extreme angulation (≥90°) proximal to or within the target lesion
7. Lesion is located in left main coronary artery
8. Thrombus in the target vessel determined by angiography or OCT
9. Subject with three-vessel disease where all three vessels require intervention
10. Additional lesion in same coronary vessel which requires treatment
11. Evidence of previous revascularization

    1. Previous PCI with or without restenosis from previous intervention
    2. Arterial or venous graft with or without lesion located within the graft or distal to a diseased arterial or saphenous vein graft Note: Lesions within 3 mm of the origin of the right coronary artery may be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1872 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) | 1 year
  It is a composite of cardiovascular death, target vessel myocardial infarction (TVMI) and clinically driven target lesion revascularization (CD TLR).

SECONDARY OUTCOMES:
Target Lesion Failure (TLF) | 30 days, 6 months, 2 years, 3 years, 4 years and 5 years
  It is a composite of cardiovascular death, target vessel myocardial infarction and clinically driven target lesion revascularization
Cardiovascular Death | 30 days, 6 months, 2 years, 3 years, 4 years and 5 years
  Defined as per the ARC-2 criteria
  The following categories will be collected:
  * Death caused by acute MI
  * Death caused by sudden cardiac arrest, including unwitnessed death
  * Death resulting from heart failure
  * Death caused by stroke
  * Death caused by cardiovascular procedures
  * Death resulting from cardiovascular hemorrhage
  * Death resulting from other cardiovascular cause.
Target Vessel Myocardial Infarction | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  * MI related to the target vessel is defined as TVMI
  * MI is defined as per the fourth universal definitions of MI
Clinically Driven Target Lesion Revascularization | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  -It is defined as repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion with following additional criteria hierarchically:
  1. Core laboratory-reported fractional flow reserve ≤0.80 or instant wave-free ratio ≤0.89
  2. Site-reported fractional flow reserve ≤0.80 or instant wave-free ratio ≤0.89
  3. Quantitative coronary analysis diameter stenosis >50% (based on the average of multiple views) with either recurrent symptoms or positive non-invasive functional test
  4. Quantitative coronary analysis diameter stenosis >70% (based on the average of multiple views) regardless of other criteria
  5. Quantitative coronary analysis diameter stenosis >70% (based on the worst view) regardless of other criteria
Target Vessel Failure | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  It is defined as the composite of cardiovascular death, target vessel myocardial infarction, and target vessel revascularization
Target Vessel Revascularization | 30 days, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  It is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel, including the target lesion revascularization
Scaffold/Stent Thrombosis Rate | : 30 days, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years
  It is defined as per ARC-2 criteria
Device Success | From the start of Index Procedure till 5 years follow ups subsequently
  It is defined as successful delivery and deployment of the study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual diameter stenosis <30% of all treated lesions as assessed by visual inspection or quantitative coronary angiography and TIMI 3 flow grade of the treated vessel
Procedure Success | From the start of Index Procedure till 5 years follow ups subsequently
  It is defined as successful delivery and deployment of the study scaffold/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual diameter stenosis <30% of all treated lesions as assessed by visual inspection or quantitative coronary angiography and TIMI 3 flow grade of the treated vessel for all target lesions without the occurrence of cardiovascular death, target vessel MI or repeat TLR during the hospital stay
Quality of Life Short Form Survey (SF-12) | Baseline, 30 days and 1 year
  Overall Health Status assessed by Short Form Survey (SF-12)